CLINICAL TRIAL: NCT07035171
Title: CABGpreHAB- Home-based Multimodal Prehabilitation (CABGpreHAB) for Elective Patients Awaiting CABG-surgery - a Feasibility Study Protocol
Brief Title: CABGpreHAB - a Feasibility Study Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Dorte Bæk Olsen, Clinical Nurse Specialist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Rigshospitalet Copenhagen
Record Dates: First submitted 2025-05-19; First posted 2025-06-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Ischaemic Heart Disease; Prehabilitation; Coronary Artery Bypass; Feasibility Studies; Multimodal Intervention; Adult
Keywords: Prehabilitation, CABG surgery, adult, preoperative,homebased
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CABGpreHAB multimodal prehabilitation intervention + usual care (Experimental): Patients randomized to the multimodal prehabilitation programme will, besides usual care, receive home-based preoperative interventions that consist of:
  Web-based exercise intervention supervised by skilled physiotherapists and delivered via a tablet. Each session lasts 60 minutes, three times per week for the prehabilitation period. Patients will be instructed to perform daily exercise tasks such as brisk walking and sit-to-stand exercises.
  Phone call and consultation delivered by a specialised nurse once a week. This consultation will deliver psychosocial support, equipping patients with coping strategies to mitigate stress, anxiety, and depression. Furthermore, nutritional advice will take place at these consultations, as well as advice on smoking cessation and alcohol cessation.
  Interventions: Other: Multimodal prehabilitation intervention
- Control group (Other): Participants assigned to the control group will receive usual care.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Multimodal prehabilitation intervention — Multimodal prehabilitation interventions (CABGpreHAB):
  * Home-based exercise intervention delivered by a skilled physiotherapist via a web-based application.
  * Nutritional intervention
  * Psycho-educative intervention
  * Smoking cessation
  * Alcohol cessation
  Arms: CABGpreHAB multimodal prehabilitation intervention + usual care
Other: Control (Standard treatment) — This includes standard information about CABG surgery, pre- and postoperative care, and postoperative physical activity advice. Patients are either admitted days before or on the day before surgery. They receive written materials and links to animated videos about preparing for surgery. This preparation includes counseling with a multidisciplinary team, including a department nurse, a physiotherapist, a cardiac anesthesiologist, and a surgeon.
  Arms: Control group

SUMMARY:
Patients with ischemic heart disease (IHD) awaiting coronary artery bypass graft (CABG) surgery often face challenges like advanced age, frailty, comorbidities, and physical inactivity. These factors, combined with the physiological and psychological stress of surgery, can hinder postoperative recovery. Traditionally, strategies to improve surgical outcomes focus on the intra- and postoperative periods. However, the pre-surgery waiting period offers a "window of opportunity" for prehabilitation, which aims to enhance patients' functional capacity through exercise, nutrition, and psychological support.

The CABGpreHAB feasibility study evaluates the feasibility of a home-based multimodal prehabilitation intervention for patients awaiting elective CABG surgery. This randomized pilot study compares the intervention plus usual care to usual care alone, assessing feasibility outcomes like recruitment, retention, attrition, fidelity, and adherence. The study aims to optimize a subsequent full-scale randomized controlled trial (RCT) and improve patient outcomes by leveraging the pre-surgery period for prehabilitation.

DETAILED DESCRIPTION:
Advanced age, frailty, comorbidity, and physical inactivity are often present in patients with ischemic heart disease (IHD) awaiting coronary artery bypass graft surgery (CABG). These characteristics, as well as the physiological impact of having surgery, are significant homeostatic disturbances where patients postoperatively suffer from physical symptoms and a lack of return to independence. Cardiac surgery invariably induces varying degrees of physiological stress, impacting multiple organ systems, and imposes a psychological burden. As age increases, patient complexity and comorbid burden grow more common in patients undergoing cardiac surgery; innovative strategies are required to alleviate the risk of adverse outcomes. Strategies to improve outcomes from surgery and accelerate return to baseline levels have traditionally focused on the intra- and postoperative period, nevertheless, the waiting period before surgery might offer an opportunity for improving the safety and outcome of the surgical intervention and improving patients' motivation in postoperative rehabilitation and recovery time. Prehabilitation is a newly introduced term that reflects a proactive process of enhancing an individual's functional capacity between diagnosis and scheduled surgery, intending to improve the patient's capacity to withstand the upcoming physiologic stress of surgery and thus avoid complications. This period of awaiting surgery is proposed as a "window of opportunity" to address poor nutritional status, low physical fitness, and high emotional distress. The role of multimodal prehabilitation combining exercise training, nutritional optimization, and psychological support, in patients with IHD awaiting CABG surgery, is sparse and unknown in a Danish setting

Objective:

This CABG preHAB feasibility study is conducted to evaluate the feasibility of delivering a homebased multimodal prehabilitation intervention for patients awaiting elective CABG surgery with the purpose to optimize a subsequent full-scale RCT.

Design:

The CABGpreHAB feasibility study is designed as a randomized pilot study, aiming to assess the feasibility of a multimodal prehabilitation intervention plus usual care versus usual care alone in patients awaiting elective CABG surgery. It is an investigator-initiated study designed as an open-label, single-center randomized controlled feasibility study (allocation ratio 1:1) with blinded outcome assessment, designed to assess the method proposed for use in a larger RCT.

Study population:

Patients aged more than 18 years awaiting elective CABG-surgery

Primary outcomes:

Feasibility outcomes include:

Recruitment and retention rates. The recruitment rate will be determined by the number of individuals participating in the study out of those who are eligible/admissible but refuse to participate. First, the investigators will evaluate the number of patients that can be included in the study during the inclusion period. A proportion of 60% or more of patients awaiting elective CABG surgery who are eligible for the study is acceptable. Retention will be assessed by the percentage of participants who remain in the study from the beginning to the end of the study (30 days post-surgery).

Attrition rates. Attrition is defined by the number of individuals who consent to participate in the study but drop out before the end of the intervention period, regardless of group allocation.

Fidelity. Fidelity of delivery of the webcam-based exercise training intervention will be assessed qualitatively by 8-10 semi-structured interviews, the day before surgery, by a research nurse.

Adherence to the interventions will be measured by using the number of telephone counselling and tele-exercise sessions delivered out of the theoretical number that could have been delivered based on the surgical wait time of each participant. Adherence to the home-based tele-exercise training sessions and telephone counselling by assessing the number of sessions applied in the intervention group. This will be collected by the patient's recorded physical activity logbook, by weekly phone calls, and by accelerometer data. Adherence with the prehabilitation program will be assessed against the target of individuals achieving > 70% of the prescribed exercise program (self-reported) + during the study follow-up with phone calls. Inclusion in the CABGpreHAB study must be attractive to at least 30% of eligible patients who meet the inclusion criteria. The interventions must be widely accepted, with at least 70% of included participants completing 70% or more of the planned sessions in the intervention group. Safety of the intervention will be determined based on the number and nature of adverse events (AE).

Secondary outcomes:

Secondary outcomes will assess the patients' responses to the multimodal prehabilitation programme, and data will be collected on explorative outcomes, measured at baseline, the day before surgery and 30 days PO.

ELIGIBILITY:
Inclusion Criteria:

* Planned to have elective isolated first-time CABG surgery.
* 18 years or older
* Two weeks or more before surgery
* Speaks and understands Danish.
* Gives written informed consent.

Exclusion Criteria:

* Patient with unstable angina pectoris and/ or MI during the last two weeks.
* Left main stem stenosis >50%
* Left ventricular ejection fraction < 35%
* Significant ventricular arrhythmia
* Orthopedic or neurologic preconditions precluding exercise training.
* Inability to attend the prehabilitation program due to physical limitations.
* Patients who have cognitive deficits that would disqualify prehabilitation.
* Severe heart failure, NYHA Class IV
* Lack of capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome: recruitement rate | Through study completition, an average of 1 year
  Determined by the number of individuals participating in the study out of those eligible during the inclusion period.
Feasibility outcome: Attrition rates | Up to 30 days post surgery index
  Defined by the numbers of individuals who give consent to participate, but drop out before study ends.
Feasibility outcome: Fidelity | preoperative
  Fidelity of delivery on the web-based exercise training intervention will be assessed qualitatively by semi-structured interviews
Feasibility outcome: Adherence rates | Preoperative
  Adherence will be assessed by measuring the number of telephone counseling and exercise sessions delivered during the intervention period.
Feasibility outcome: Safety | From enrolement to the day before surgery
  Safety of the intervention will be determined based on the number and nature of adverse events.

SECONDARY OUTCOMES:
Exercise capacity | Three times: at baseline, preoperative and 30 days post surgery index
  6MWT measures total walking distance in meters completed in six minutes
Muscle strength | Three times: at baseline, preoperative and 30 days post surgery index
  30 seconds sit-to-stand measured by numbers of sit-to-stands in 30 seconds
Muscle strength handgrip | At baseline and preoperative
  Measured in kilograms using a hand-held dynamometer
Bodycomposition | At baseline and preoperative
  Using a Bioelectrical Impedance Analyzer (BIA), body composition estimation:
  fat mass in kilograms,
  Fat mass as a percentage of weight,
  Fat-free mass in kilograms,
  Fat-free mass as a percentage of weight
Nutritional status | At baseline and preoperative
  Weight and height combined to report BMI in kg/m^2,
  and
  Screened by the NRS2002 score
Daily physical activity | Three times: at baseline, preoperative and 30 days post surgery index
  SENS motion accelerometer measures minutes of physical activity as
  steps, Cyckling running Standing Laying
HRQOL | Three times: at baseline, preoperative and 30 days post surgery index
  The Questionnaire SF-12 measures overall health status
Heart-specific QoL | Three times: at baseline, preoperative and 30 days post surgery index
  The Questionnaire HeartQoL measures health-related quality of life in patients with ischemic heart disease
Anxiety | Three times: at baseline, preoperative and 30 days post surgery index
  The State-Trait Anxiety Inventory Questionnaire measures two disitnc types of anxiety
Depression | Three times: at baseline, preoperative and 30 days post surgery index
  The PHQ-4 Questionnaire measures depression and anxiety
Sense of coherence | At baseline
  The SOC-13 Questionnaire assesses an individual´s ability to manage stress and maintain health
Self-efficacy/self-management | Three times: at baseline, preoperative and 30 days post surgery index
  The PAM13 Questionnaire assesses an individual's knowledge, skill, and confidence for self-management
Tobacco uses status | Three times: at baseline, preoperative and 30 days post surgery index
  Self-Reported Questionnaire
Alcohol uses status | Three times: at baseline, preoperative and 30 days post surgery index
  Self-Reported Questionnaire

OTHER OUTCOMES:
Complications postoperatively | From date of surgery and up to 30 days postopetively.
  Rates of pneumonia, atelectasis, hemorrhage, cardiac arrhythmias, and delirium will be measured postoperatively
ICU-LOS | From date and time of surgery until the date and time of discharge to the ward.
  ICU-LOS will be calculated in hours
LOS | From date of surgery until date of discharge from the ward
  LOS will be calculated in days
DAOH30 | From date of surgery and up to 30 days postopetively.
  DAOH30 will be calculated in days
Participating in Cardiac rehabilitation | At 30 days postoperatively
  Participation will be calculated in percentage
Bloodtest | At baseline and postoperatively day 4
  HGB measured in mmol/l Albumin measured in g/l CRP measured in mg/l Creatinine measured in micromol/l

CONTACTS AND LOCATIONS:
Overall Officials: Ida E Hoejskov, PhD, Principal Investigator — Department of Heart Disease, Rigshospitalet, Copenhagen University Hospital
Locations (1):
- The Department of Heart and Lung Surgery, Copenhagen University hospital Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT07035171/Prot_000.pdf